CLINICAL TRIAL: NCT04908592
Title: Efficacy of Dexamethasone in Attenuation of Postinduction Hypotension in Geriatric Patients Undergoing General Anesthesia: a Randomized Controlled Trial
Brief Title: Efficacy of Dexamethasone in Attenuation of Postinduction Hypotension in Geriatric Patients Undergoing General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 289/ 2021
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D Group (50 patients) (Active Comparator)
  Interventions: Drug: Dexamethasone
- C Group (50 patients) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive dexamethasone 8 mg diluted in 100 ml 0.9% normal saline (NS) IVI over 15 min 2 h preoperatively.
  Arms: D Group (50 patients)
Other: Placebo — Patients will receive 100 ml 0.9% normal saline (NS) IVI over 15 min 2 h preoperatively.
  Arms: C Group (50 patients)

SUMMARY:
* Geriatric patients who undergo general anesthesia experience post induction hypotension which is treated with intravenous fluids and ephedrine. The main cause of post-induction hypotension is the decrease in the sympathetic outflow causing arterial vasodilatation, a decrease in venous return and consequently the activation of the Bezold Jarish reflex (BJR) that elicits a triad of bradycardia, vasodilatation and further hypotension. BJR is elicited by activation of 5-HT3 receptors within the intracardiac vagal nerve endings.
* Glucocorticoids in general inhibit 5-HT3 expression and dexamethasone was found to decrease the level of 5-HT3 in the cerebral cortex and hippocampus in developing rats. So, the research team hypothesizes that dexamethasone can attenuate the postinduction hypotension in geriatric patients undergoing general anesthesia if administered preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Physical Status Class-I and II.
2. Elective surgery under general anesthesia.

Exclusion Criteria:

1. Emergency surgeries.
2. Ischemic heart disease.
3. Peptic ulcer & active infection.
4. Psychiatric disorder.
5. Patients on steroids or serotonin related medications (e.g., selective serotonin reuptake inhibitor).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with hypotension (25% decrease below the baseline for mean blood pressure (mmHg). | intraoperative
  The proportion of patients with hypotension (25% decrease below the baseline for mean blood pressure (mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No